CLINICAL TRIAL: NCT05001100
Title: A Rehabilitation With Virtual Reality in Patients After Hip Arthroplasty Surgery (VRRS2018)
Acronym: VRRS2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRRS2018
Record Dates: First submitted 2021-07-29; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Hip Disease
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional rehabilitation (Active Comparator): 32 subjects will undergo a virtual motor-reality training during the post-surgical rehabilitation period with VRSS
  Interventions: Other: rehabilitation
- Rehabilitation with virtual reality (Experimental): 32 subjects with demographic characteristics similar to the subjects of the Vrrs arm will undergo the habitual rehabilitative physiotherapy.
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — rehabilitation

SUMMARY:
.Assessing efficacy of rehabilitation with virtual reality exercises compared to traditional rehabilitation in the patient's operated hip arthroplasty

DETAILED DESCRIPTION:
Randomized controlled clinical study: Comparison of clinical efficacy between rehabilitation with virtual reality (VRRS) and traditional physiotherapy in post-surgical rehabilitation treatment in hospital. Motor clinical evaluations will be carried out in both groups.

Vrrs Arm: 32 subjects will undergo a virtual motor-reality training during the post-surgical rehabilitation period.

Physiotherapist's arm: 32 subjects with demographic characteristics similar to the subjects of the Vrrs arm will undergo the habitual rehabilitative physiotherapy.

According to normal clinical practice, both groups perform a co-intervention in addition to the assigned group; Manual therapy with exercises and functional activity (walk and stairs).

ELIGIBILITY:
Inclusion Criteria:

- hip arthroplasty

Exclusion Criteria:

* patient with resence of neurological and psychiatric disorders
* minor patient

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-11-07 (Actual)

PRIMARY OUTCOMES:
disability measurement | on the 21st day
  WOMAC (Western Ontario and McMaster University) Osteoarthritis index

SECONDARY OUTCOMES:
pain measurement | on the 10st day
  visual analoge scale VAS

CONTACTS AND LOCATIONS:
Overall Officials: cristina beretta, MD, Principal Investigator — istituto galeazzi
Locations (1):
- Irccs Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No